CLINICAL TRIAL: NCT00755677
Title: Exploring the Health Benefits Associated With Daily Pulse Consumption in Individuals With Peripheral Arterial Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Boniface Hospital (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr.Peter Zahradka, Professor, Department of Physiology, St. Boniface Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pulse Study
Record Dates: First submitted 2008-09-11; First posted 2008-09-19 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Pulse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pulses (Other): Interventional. Participants are registered sequentially to undergo daily consumption of pulses for eight weeks
  Interventions: Other: Pulses

INTERVENTIONS:
Other: Pulses — subjects consume 1 pulse food daily for eight weeks

SUMMARY:
This is a single site, open registration, dietary proof of concept, food substance study designed to explore the health benefits associated with daily pulse consumption in individuals with peripheral arterial disease. The investigators hypothesis that a diet containing at least one serving of pulse crops (dried beans, peas, lentil, chickpeas) per day provides flavonoid compounds that improve cardiovascular health by increasing the levels of serum adiponectin is based on evidence from the literature that indicates flavonoids present in these foods are capable of improving arterial stiffness and reducing hypercholesterolemia.

DETAILED DESCRIPTION:
Objectives:

* Correlate serum adiponectin levels with daily intake of pulses in individuals with peripheral arterial disease
* Monitor changes in arterial stiffness and endothelial dysfunction in individuals with early stage cardiovascular disease
* Determine the tolerability of daily consumption of pulses in the targeted population
* Identify changes in the expression profile of white blood cells.

Study Duration: 12 months

Study Design:

* This is a single site, open registration, dietary proof of concept, food substance study designed to explore the health benefits associated with daily pulse consumption in individuals with arterial disease
* Each subject will undergo a 7-day adaptation period consisting of a consumption of ¼ cup of pulses per serving daily, followed by a minimum of ½ cup of pulses per serving daily
* Total duration of subject participation is 8 weeks;
* Subjects will be asked to attend 3 in-person clinic visits over the duration of their participation in the study for screening, registration/baseline and end of study assessments
* Telephone follow-up to subjects will occur at weeks 1,2,4, and 6
* Both clinical assessment and subject-based data will be collected at various points of the study schedule
* Subjects will be asked to complete a food frequency questionnaire at the outset, maintain a 3-day food record at two separate occasions, and undergo a brief semi-structured interview during the telephone follow-up assessments of the study

Assessments:

1. Screening Visit: Informed consent; inclusion/exclusion criteria assessment; medical history; physical exam; food frequency questionnaire; 3-day food record
2. Registration/Baseline: Registration; assess for changes to medical history (including medication profile) and physical condition; urine sample; fasting blood sample; assessment of arterial stiffness and ankle-brachial index; begin adaptation period (7 days)with food items containing ¼ c of pulses per serving
3. Visits 1,2,4 & 6: Telephone follow-up to assess adverse events and tolerability with semi-structured subject interview; distribution (weekly) of food items containing a minimum of ½ cup pulses per serving; 3-day food record repeated at week 6
4. Visit 8 (final): Assess for adverse events and changes to medical history and physical exam; urine sample; fasting blood sample collection; assessment of arterial stiffness and and ankle-brachial index

Outcomes:

* Descriptive analysis of clinical data: Demographics, medical history, physical findings, concomitant medications and adverse events
* Identification of changes in endothelial function (determined by measuring pulse wave velocity (PWV), ankle-brachial index, soluble adhesion molecule levels and coagulation status) in response to dietary modification
* Correlation of serum adiponectin levels, including adiponectin multimers and truncated form (globular adiponectin) with endothelial function
* Correlation of changes in endothelial cell function with serum isoflavone levels
* Qualitative analysis of data collected from semi-structured subject interviews to assess parameters associated with tolerability of diet and to identify favoured recipes
* Profile cohort using 55,000 gene microarray to identify potential biomarkers and changes in gene expression (phenotype mapping) induced by diet
* Use microarrays to examine gene methylation and single nucleotide polymorphisms (SNP) in DNA samples to determine if changes in expression profile are due to epigenetic modification (global) or allelic (individual) variation in the study cohort in response to a pulse-enriched diet
* Serum and urinary eicosanoids will be analyzed by a multi-step procedure utilizing liquid chromatography, derivitization steps, thin-layer chromatography and gas chromatography-mass spectrometry
* Serum will also be analyzed for fatty acid composition using thin-layer chromatography and gas chromatography

ELIGIBILITY:
Inclusion Criteria:

* Presence of peripheral arterial disease including those with claudication as defined by an ankle brachial index of ≤ 0.90 and asymptomatic carotid stenosis lesion of > 50%
* Male or female (> 40 years of age)
* Willing to comply with the protocol requirements
* Willing to provide informed consent
* Stable medication profile with no changes anticipated for the duration of the proposed study schedule (8 weeks)

Exclusion Criteria:

* Renal failure requiring dialysis
* Currently smoking
* Hormone replacement therapy
* Inability to adhere to a regular diet
* Additional intake of pulses outside the planned daily requirements outlined in the study
* History of gastrointestinal reactions or allergies to pulses

Ages: 40 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-03; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Identification of changes in endothelial function in response to dietary modification | baseline, week 8
Correlation of serum adiponectin levels | baseline, week 8
Correlation of changes in endothelial cell function with serum isoflavone levels | baseline, week 8
Genetic Profiling | baseline, week 8
Analysis of serum and urinary eicosanoids | baseline, week 8
Serum analysis for fatty acid composition | baseline, week 8

SECONDARY OUTCOMES:
Descriptive analysis of clinical data: Demographics, medical history, | baseline
Physical findings, concomitant medications and adverse events | baseline, weekly for 8 weeks
Qualitative analysis of data collected from semi-structured subject interviews | week 1, week 2, week 4, week 6, week 8
(Compliance/tolerability/side effects) | week 1, week 2, week 4, week 6, week 8

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zahradka, PhD, Principal Investigator — St. Boniface Hospital
Locations (1):
- St. Boniface General Hospital, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Wilson PW, D'Agostino RB, Sullivan L, Parise H, Kannel WB. Overweight and obesity as determinants of cardiovascular risk: the Framingham experience. Arch Intern Med. 2002 Sep 9;162(16):1867-72. doi: 10.1001/archinte.162.16.1867. PMID 12196085
- [Background] Calkin AC, Allen TJ. Diabetes mellitus-associated atherosclerosis: mechanisms involved and potential for pharmacological invention. Am J Cardiovasc Drugs. 2006;6(1):15-40. doi: 10.2165/00129784-200606010-00003. PMID 16489846
- [Background] Juvenile Diabetes Research Foundation (2005) http://www jdrf org au/publications/factsheets/complications html
- [Background] Li TY, Rana JS, Manson JE, Willett WC, Stampfer MJ, Colditz GA, Rexrode KM, Hu FB. Obesity as compared with physical activity in predicting risk of coronary heart disease in women. Circulation. 2006 Jan 31;113(4):499-506. doi: 10.1161/CIRCULATIONAHA.105.574087. PMID 16449729
- [Background] British Heart Foundation Statistics (2006) www heartstats org
- [Background] Houston DK, Stevens J, Cai J, Haines PS. Dairy, fruit, and vegetable intakes and functional limitations and disability in a biracial cohort: the Atherosclerosis Risk in Communities Study. Am J Clin Nutr. 2005 Feb;81(2):515-22. doi: 10.1093/ajcn.81.2.515. PMID 15699243
- [Background] Hu FB, Willett WC. Optimal diets for prevention of coronary heart disease. JAMA. 2002 Nov 27;288(20):2569-78. doi: 10.1001/jama.288.20.2569. PMID 12444864
- [Background] Bazzano LA, Serdula MK, Liu S. Dietary intake of fruits and vegetables and risk of cardiovascular disease. Curr Atheroscler Rep. 2003 Nov;5(6):492-9. doi: 10.1007/s11883-003-0040-z. PMID 14525683
- [Background] Anderson JW, Major AW. Pulses and lipaemia, short- and long-term effect: potential in the prevention of cardiovascular disease. Br J Nutr. 2002 Dec;88 Suppl 3:S263-71. doi: 10.1079/BJN2002716. PMID 12498626
- [Background] Castro IA, Barroso LP, Sinnecker P. Functional foods for coronary heart disease risk reduction: a meta-analysis using a multivariate approach. Am J Clin Nutr. 2005 Jul;82(1):32-40. doi: 10.1093/ajcn.82.1.32. PMID 16002797
- [Background] Rowland I. Optimal nutrition: fibre and phytochemicals. Proc Nutr Soc. 1999 May;58(2):415-9. doi: 10.1017/s0029665199000543. PMID 10466185
- [Background] Gylling H, Miettinen TA. The effect of plant stanol- and sterol-enriched foods on lipid metabolism, serum lipids and coronary heart disease. Ann Clin Biochem. 2005 Jul;42(Pt 4):254-63. doi: 10.1258/0004563054255605. PMID 15989725
- [Background] Hertog MG, Feskens EJ, Hollman PC, Katan MB, Kromhout D. Dietary antioxidant flavonoids and risk of coronary heart disease: the Zutphen Elderly Study. Lancet. 1993 Oct 23;342(8878):1007-11. doi: 10.1016/0140-6736(93)92876-u. PMID 8105262
- [Background] Keli SO, Hertog MG, Feskens EJ, Kromhout D. Dietary flavonoids, antioxidant vitamins, and incidence of stroke: the Zutphen study. Arch Intern Med. 1996 Mar 25;156(6):637-42. PMID 8629875
- [Background] Wylie-Rosett J, Segal-Isaacson CJ, Segal-Isaacson A. Carbohydrates and increases in obesity: does the type of carbohydrate make a difference? Obes Res. 2004 Nov;12 Suppl 2:124S-9S. doi: 10.1038/oby.2004.277. PMID 15601960
- [Background] Delzenne NM, Cani PD. A place for dietary fibre in the management of the metabolic syndrome. Curr Opin Clin Nutr Metab Care. 2005 Nov;8(6):636-40. doi: 10.1097/01.mco.0000171124.06408.71. PMID 16205465
- [Background] Matvienko OA, Lewis DS, Swanson M, Arndt B, Rainwater DL, Stewart J, Alekel DL. A single daily dose of soybean phytosterols in ground beef decreases serum total cholesterol and LDL cholesterol in young, mildly hypercholesterolemic men. Am J Clin Nutr. 2002 Jul;76(1):57-64. doi: 10.1093/ajcn/76.1.57. PMID 12081816
- [Background] Sharma RD. Isoflavones and hypercholesterolemia in rats. Lipids. 1979 Jun;14(6):535-9. doi: 10.1007/BF02533528. PMID 459719
- [Background] Beninger CW, Hosfield GL. Antioxidant activity of extracts, condensed tannin fractions, and pure flavonoids from Phaseolus vulgaris L. seed coat color genotypes. J Agric Food Chem. 2003 Dec 31;51(27):7879-83. doi: 10.1021/jf0304324. PMID 14690368
- [Background] Tsuda T, Ueno Y, Aoki H, Koda T, Horio F, Takahashi N, Kawada T, Osawa T. Anthocyanin enhances adipocytokine secretion and adipocyte-specific gene expression in isolated rat adipocytes. Biochem Biophys Res Commun. 2004 Mar 26;316(1):149-57. doi: 10.1016/j.bbrc.2004.02.031. PMID 15003523
- [Background] Cassidy A, Brown JE, Hawdon A, Faughnan MS, King LJ, Millward J, Zimmer-Nechemias L, Wolfe B, Setchell KD. Factors affecting the bioavailability of soy isoflavones in humans after ingestion of physiologically relevant levels from different soy foods. J Nutr. 2006 Jan;136(1):45-51. doi: 10.1093/jn/136.1.45. PMID 16365057
- [Background] Milerova J, Cerovska J, Zamrazil V, Bilek R, Lapcik O, Hampl R. Actual levels of soy phytoestrogens in children correlate with thyroid laboratory parameters. Clin Chem Lab Med. 2006;44(2):171-4. doi: 10.1515/CCLM.2006.031. PMID 16475902
- [Background] Huang Y, Cao S, Nagamani M, Anderson KE, Grady JJ, Lu LJ. Decreased circulating levels of tumor necrosis factor-alpha in postmenopausal women during consumption of soy-containing isoflavones. J Clin Endocrinol Metab. 2005 Jul;90(7):3956-62. doi: 10.1210/jc.2005-0161. Epub 2005 Apr 19. PMID 15840745
- [Background] Colacurci N, Chiantera A, Fornaro F, de Novellis V, Manzella D, Arciello A, Chiantera V, Improta L, Paolisso G. Effects of soy isoflavones on endothelial function in healthy postmenopausal women. Menopause. 2005 May-Jun;12(3):299-307. doi: 10.1097/01.gme.0000147017.23173.5b. PMID 15879919
- [Background] Heald CL, Bolton-Smith C, Ritchie MR, Morton MS, Alexander FE. Phyto-oestrogen intake in Scottish men: use of serum to validate a self-administered food-frequency questionnaire in older men. Eur J Clin Nutr. 2006 Jan;60(1):129-35. doi: 10.1038/sj.ejcn.1602277. PMID 16205743
- [Background] Ozasa K, Nakao M, Watanabe Y, Hayashi K, Miki T, Mikami K, Mori M, Sakauchi F, Washio M, Ito Y, Suzuki K, Kubo T, Wakai K, Tamakoshi A; JACC Study Group. Association of serum phytoestrogen concentration and dietary habits in a sample set of the JACC Study. J Epidemiol. 2005 Jun;15 Suppl 2(Suppl II):S196-202. doi: 10.2188/jea.15.s196. PMID 16127234
- [Background] Ma Y, Chiriboga D, Olendzki BC, Nicolosi R, Merriam PA, Ockene IS. Effect of soy protein containing isoflavones on blood lipids in moderately hypercholesterolemic adults: a randomized controlled trial. J Am Coll Nutr. 2005 Aug;24(4):275-85. doi: 10.1080/07315724.2005.10719475. PMID 16093405
- [Background] Trayhurn P, Bing C, Wood IS. Adipose tissue and adipokines--energy regulation from the human perspective. J Nutr. 2006 Jul;136(7 Suppl):1935S-1939S. doi: 10.1093/jn/136.7.1935S. PMID 16772463
- [Background] Kelesidis T, Mantzoros CS. The emerging role of leptin in humans. Pediatr Endocrinol Rev. 2006 Mar;3(3):239-48. PMID 16639389
- [Background] Beltowski J. Leptin and atherosclerosis. Atherosclerosis. 2006 Nov;189(1):47-60. doi: 10.1016/j.atherosclerosis.2006.03.003. Epub 2006 Apr 3. PMID 16580676
- [Background] Haluzik M, Haluzikova D. The role of resistin in obesity-induced insulin resistance. Curr Opin Investig Drugs. 2006 Apr;7(4):306-11. PMID 16625816
- [Background] Lam KS, Xu A. Adiponectin: protection of the endothelium. Curr Diab Rep. 2005 Aug;5(4):254-9. doi: 10.1007/s11892-005-0019-y. PMID 16033674
- [Background] Do D, Alvarez J, Chiquette E, Chilton R. The good fat hormone: adiponectin and cardiovascular disease. Curr Atheroscler Rep. 2006 Mar;8(2):94-9. doi: 10.1007/s11883-006-0045-5. PMID 16510042
- [Background] Haluzik M. Adiponectin and its potential in the treatment of obesity, diabetes and insulin resistance. Curr Opin Investig Drugs. 2005 Oct;6(10):988-93. PMID 16259219
- [Background] Okamoto Y, Kihara S, Ouchi N, Nishida M, Arita Y, Kumada M, Ohashi K, Sakai N, Shimomura I, Kobayashi H, Terasaka N, Inaba T, Funahashi T, Matsuzawa Y. Adiponectin reduces atherosclerosis in apolipoprotein E-deficient mice. Circulation. 2002 Nov 26;106(22):2767-70. doi: 10.1161/01.cir.0000042707.50032.19. PMID 12451000
- [Background] Clasen R, Schupp M, Foryst-Ludwig A, Sprang C, Clemenz M, Krikov M, Thone-Reineke C, Unger T, Kintscher U. PPARgamma-activating angiotensin type-1 receptor blockers induce adiponectin. Hypertension. 2005 Jul;46(1):137-43. doi: 10.1161/01.HYP.0000168046.19884.6a. Epub 2005 Jun 6. PMID 15939809
- [Background] Murdolo G, Smith U. The dysregulated adipose tissue: a connecting link between insulin resistance, type 2 diabetes mellitus and atherosclerosis. Nutr Metab Cardiovasc Dis. 2006 Mar;16 Suppl 1:S35-8. doi: 10.1016/j.numecd.2005.10.016. Epub 2006 Feb 9. PMID 16530128
- [Background] Smith J, Al-Amri M, Dorairaj P, Sniderman A. The adipocyte life cycle hypothesis. Clin Sci (Lond). 2006 Jan;110(1):1-9. doi: 10.1042/CS20050110. PMID 16336200
- [Background] Lofgren P, Andersson I, Wahrenberg H, Hoffstedt J. No difference in lipolysis or glucose transport of subcutaneous fat cells between moderate-fat and low-fat hypocaloric diets in obese women. Horm Metab Res. 2005 Dec;37(12):734-40. doi: 10.1055/s-2005-921095. PMID 16372226
- [Background] Farnier C, Krief S, Blache M, Diot-Dupuy F, Mory G, Ferre P, Bazin R. Adipocyte functions are modulated by cell size change: potential involvement of an integrin/ERK signalling pathway. Int J Obes Relat Metab Disord. 2003 Oct;27(10):1178-86. doi: 10.1038/sj.ijo.0802399. PMID 14513065
- [Background] Bays H, Dujovne CA. Adiposopathy is a more rational treatment target for metabolic disease than obesity alone. Curr Atheroscler Rep. 2006 Mar;8(2):144-56. doi: 10.1007/s11883-006-0052-6. PMID 16510049
- [Background] Wu ZH, Zhao SP. Adipocyte: a potential target for the treatment of atherosclerosis. Med Hypotheses. 2006;67(1):82-6. doi: 10.1016/j.mehy.2005.12.042. Epub 2006 Feb 24. PMID 16500036
- [Background] Erol A. The role of fat tissue in the cholesterol lowering and the pleiotropic effects of statins--statins activate the generation of metabolically more capable adipocytes. Med Hypotheses. 2005;64(1):69-73. doi: 10.1016/j.mehy.2004.06.014. PMID 15533614
- [Background] Noto A, Zahradka P, Yurkova N, Xie X, Nitschmann E, Ogborn M, Taylor CG. Conjugated linoleic acid reduces hepatic steatosis, improves liver function, and favorably modifies lipid metabolism in obese insulin-resistant rats. Lipids. 2006 Feb;41(2):179-88. doi: 10.1007/s11745-006-5086-6. PMID 17707984
- [Background] Dzau VJ, Braun-Dullaeus RC, Sedding DG. Vascular proliferation and atherosclerosis: new perspectives and therapeutic strategies. Nat Med. 2002 Nov;8(11):1249-56. doi: 10.1038/nm1102-1249. No abstract available. PMID 12411952
- [Background] Leterme P. Recommendations by health organizations for pulse consumption. Br J Nutr. 2002 Dec;88 Suppl 3:S239-42. doi: 10.1079/BJN2002712. PMID 12498622
- [Background] Statpub (2004) World edible bean industry growing slowly. http://www statpub com/open/123607/html
- [Background] van der Vleuten GM, van Tits LJ, den Heijer M, Lemmers H, Stalenhoef AF, de Graaf J. Decreased adiponectin levels in familial combined hyperlipidemia patients contribute to the atherogenic lipid profile. J Lipid Res. 2005 Nov;46(11):2398-404. doi: 10.1194/jlr.M500212-JLR200. Epub 2005 Aug 16. PMID 16106049
- [Background] Yoshida H, Hirowatari Y, Kurosawa H, Tada N. Implications of decreased serum adiponectin for type IIb hyperlipidaemia and increased cholesterol levels of very-low-density lipoprotein in type II diabetic patients. Clin Sci (Lond). 2005 Sep;109(3):297-302. doi: 10.1042/CS20040353. PMID 15907189
- [Background] Anderson TJ. Arterial stiffness or endothelial dysfunction as a surrogate marker of vascular risk. Can J Cardiol. 2006 Feb;22 Suppl B(Suppl B):72B-80B. doi: 10.1016/s0828-282x(06)70990-4. PMID 16498516
- [Background] Tuomisto TT, Binder BR, Yla-Herttuala S. Genetics, genomics and proteomics in atherosclerosis research. Ann Med. 2005;37(5):323-32. doi: 10.1080/07853890510011949. PMID 16179268
- [Background] Guillon F, Champ MM. Carbohydrate fractions of legumes: uses in human nutrition and potential for health. Br J Nutr. 2002 Dec;88 Suppl 3:S293-306. doi: 10.1079/BJN2002720. PMID 12498630
- [Background] Rizkalla SW, Bellisle F, Slama G. Health benefits of low glycaemic index foods, such as pulses, in diabetic patients and healthy individuals. Br J Nutr. 2002 Dec;88 Suppl 3:S255-62. doi: 10.1079/BJN2002715. PMID 12498625
- [Background] Pittaway JK, Ahuja KD, Chronopoulos A et al (2004) The effect of chickpeas on human serum lipids and lipoproteins. Asia Pac J Clin Nutr 13: S70-S75.
- [Background] He XZ, Reddy JT, Dixon RA. Stress responses in alfalfa (Medicago sativa L). XXII. cDNA cloning and characterization of an elicitor-inducible isoflavone 7-O-methyltransferase. Plant Mol Biol. 1998 Jan;36(1):43-54. doi: 10.1023/a:1005938121453. PMID 9484461
- [Background] Sumner LW, Paiva NL, Dixon RA, Geno PW. High-performance liquid chromatography/continuous-flow liquid secondary ion mass spectrometry of flavonoid glycosides in leguminous plant extracts. J Mass Spectrom. 1996 May;31(5):472-85. doi: 10.1002/(SICI)1096-9888(199605)31:53.0.CO;2-E. PMID 8799289
- [Background] Teede HJ, McGrath BP, DeSilva L, Cehun M, Fassoulakis A, Nestel PJ. Isoflavones reduce arterial stiffness: a placebo-controlled study in men and postmenopausal women. Arterioscler Thromb Vasc Biol. 2003 Jun 1;23(6):1066-71. doi: 10.1161/01.ATV.0000072967.97296.4A. Epub 2003 Apr 24. PMID 12714433
- [Background] DiCenzo GL, VanEtten HD. Studies on the late steps of (+) pisatin biosynthesis: evidence for (-) enantiomeric intermediates. Phytochemistry. 2006 Apr;67(7):675-83. doi: 10.1016/j.phytochem.2005.12.027. Epub 2006 Feb 28. PMID 16504226
- [Background] Tiemann K, Inze D, Van Montagu M, Barz W. Pterocarpan phytoalexin biosynthesis in elicitor-challenged chickpea (Cicer arietinum L.) cell cultures. Purification, characterization and cDNA cloning of NADPH:isoflavone oxidoreductase. Eur J Biochem. 1991 Sep 15;200(3):751-7. doi: 10.1111/j.1432-1033.1991.tb16241.x. PMID 1915347
- [Background] Robbins MP, Bolwell GP, Dixon RA. Metabolic changes in elicitor-treated bean cells. Selectivity of enzyme induction in relation to phytoalexin accumulation. Eur J Biochem. 1985 May 2;148(3):563-9. doi: 10.1111/j.1432-1033.1985.tb08877.x. PMID 3996394
- [Background] Ohkawara S, Okuma Y, Uehara T, Yamagishi T, Nomura Y. Astrapterocarpan isolated from Astragalus membranaceus inhibits proliferation of vascular smooth muscle cells. Eur J Pharmacol. 2005 Nov 21;525(1-3):41-7. doi: 10.1016/j.ejphar.2005.08.063. Epub 2005 Nov 16. PMID 16297381
- [Background] Genest J, Frohlich J, Fodor G, McPherson R; Working Group on Hypercholesterolemia and Other Dyslipidemias. Recommendations for the management of dyslipidemia and the prevention of cardiovascular disease: summary of the 2003 update. CMAJ. 2003 Oct 28;169(9):921-4. No abstract available. PMID 14581310
- [Background] Williamson G, Manach C. Bioavailability and bioefficacy of polyphenols in humans. II. Review of 93 intervention studies. Am J Clin Nutr. 2005 Jan;81(1 Suppl):243S-255S. doi: 10.1093/ajcn/81.1.243S. PMID 15640487
- [Background] Yamauchi T, Kamon J, Waki H, Imai Y, Shimozawa N, Hioki K, Uchida S, Ito Y, Takakuwa K, Matsui J, Takata M, Eto K, Terauchi Y, Komeda K, Tsunoda M, Murakami K, Ohnishi Y, Naitoh T, Yamamura K, Ueyama Y, Froguel P, Kimura S, Nagai R, Kadowaki T. Globular adiponectin protected ob/ob mice from diabetes and ApoE-deficient mice from atherosclerosis. J Biol Chem. 2003 Jan 24;278(4):2461-8. doi: 10.1074/jbc.M209033200. Epub 2002 Nov 12. PMID 12431986
- [Background] Tsao TS, Tomas E, Murrey HE, Hug C, Lee DH, Ruderman NB, Heuser JE, Lodish HF. Role of disulfide bonds in Acrp30/adiponectin structure and signaling specificity. Different oligomers activate different signal transduction pathways. J Biol Chem. 2003 Dec 12;278(50):50810-7. doi: 10.1074/jbc.M309469200. Epub 2003 Sep 30. PMID 14522956
- [Background] Boisclair MD, Ireland H, Lane DA. Assessment of hypercoagulable states by measurement of activation fragments and peptides. Blood Rev. 1990 Mar;4(1):25-40. doi: 10.1016/0268-960x(90)90014-j. PMID 2182146
- [Background] Wang G, Woo CW, Sung FL, Siow YL, O K. Increased monocyte adhesion to aortic endothelium in rats with hyperhomocysteinemia: role of chemokine and adhesion molecules. Arterioscler Thromb Vasc Biol. 2002 Nov 1;22(11):1777-83. doi: 10.1161/01.atv.0000035404.18281.37. PMID 12426204
- [Background] Barnes S, Coward L, Kirk M, Sfakianos J. HPLC-mass spectrometry analysis of isoflavones. Proc Soc Exp Biol Med. 1998 Mar;217(3):254-62. doi: 10.3181/00379727-217-44230. PMID 9492333
- [Background] Oliver JJ, Webb DJ. Noninvasive assessment of arterial stiffness and risk of atherosclerotic events. Arterioscler Thromb Vasc Biol. 2003 Apr 1;23(4):554-66. doi: 10.1161/01.ATV.0000060460.52916.D6. Epub 2003 Feb 6. PMID 12615661
- [Background] Celotti F, Durand T. The metabolic effects of inhibitors of 5-lipoxygenase and of cyclooxygenase 1 and 2 are an advancement in the efficacy and safety of anti-inflammatory therapy. Prostaglandins Other Lipid Mediat. 2003 Jul;71(3-4):147-62. doi: 10.1016/s1098-8823(03)00039-x. PMID 14518558
- [Background] Brune K. Safety of anti-inflammatory treatment--new ways of thinking. Rheumatology (Oxford). 2004 Feb;43 Suppl 1:i16-20. doi: 10.1093/rheumatology/keh104. PMID 14752171
- [Background] de Gaetano G, Donati MB, Cerletti C. Prevention of thrombosis and vascular inflammation: benefits and limitations of selective or combined COX-1, COX-2 and 5-LOX inhibitors. Trends Pharmacol Sci. 2003 May;24(5):245-52. doi: 10.1016/S0165-6147(03)00077-4. PMID 12767724
- [Background] Fischer S, Weber PC. Thromboxane (TX)A3 and prostaglandin (PG)I3 are formed in man after dietary eicosapentaenoic acid: identification and quantification by capillary gas chromatography-electron impact mass spectrometry. Biomed Mass Spectrom. 1985 Sep;12(9):470-6. doi: 10.1002/bms.1200120905. PMID 2996649
- [Background] Rupp H, Turcani M, Ohkubo T, Maisch B, Brilla CG. Dietary linolenic acid-mediated increase in vascular prostacyclin formation. Mol Cell Biochem. 1996 Sep 6;162(1):59-64. doi: 10.1007/BF00250996. PMID 8905626
- [Background] Kabagambe EK, Baylin A, Ruiz-Narvarez E, Siles X, Campos H. Decreased consumption of dried mature beans is positively associated with urbanization and nonfatal acute myocardial infarction. J Nutr. 2005 Jul;135(7):1770-5. doi: 10.1093/jn/135.7.1770. PMID 15987863
- [Background] Franke AA, Custer LJ, Cerna CM, Narala K. Rapid HPLC analysis of dietary phytoestrogens from legumes and from human urine. Proc Soc Exp Biol Med. 1995 Jan;208(1):18-26. doi: 10.3181/00379727-208-43826. PMID 7892289
- [Background] Renard C, Van Obberghen E. Role of diabetes in atherosclerotic pathogenesis. What have we learned from animal models? Diabetes Metab. 2006 Feb;32(1):15-29. doi: 10.1016/s1262-3636(07)70243-4. PMID 16523183
- [Background] Yamagishi S, Imaizumi T. Diabetic vascular complications: pathophysiology, biochemical basis and potential therapeutic strategy. Curr Pharm Des. 2005;11(18):2279-99. doi: 10.2174/1381612054367300. PMID 16022668
- [Background] Okada K, Maeda N, Kikuchi K, Tatsukawa M, Sawayama Y, Hayashi J. Pravastatin improves insulin resistance in dyslipidemic patients. J Atheroscler Thromb. 2005;12(6):322-9. doi: 10.5551/jat.12.322. PMID 16394616
- [Background] Lamendola C, Abbasi F, Chu JW, Hutchinson H, Cain V, Leary E, McLaughlin T, Stein E, Reaven G. Comparative effects of rosuvastatin and gemfibrozil on glucose, insulin, and lipid metabolism in insulin-resistant, nondiabetic patients with combined dyslipidemia. Am J Cardiol. 2005 Jan 15;95(2):189-93. doi: 10.1016/j.amjcard.2004.09.005. PMID 15642550
- [Background] Beckman JA, Creager MA. The nonlipid effects of statins on endothelial function. Trends Cardiovasc Med. 2006 Jul;16(5):156-62. doi: 10.1016/j.tcm.2006.03.003. PMID 16781949
- [Background] Fichtlscherer S, Schmidt-Lucke C, Bojunga S, Rossig L, Heeschen C, Dimmeler S, Zeiher AM. Differential effects of short-term lipid lowering with ezetimibe and statins on endothelial function in patients with CAD: clinical evidence for 'pleiotropic' functions of statin therapy. Eur Heart J. 2006 May;27(10):1182-90. doi: 10.1093/eurheartj/ehi881. Epub 2006 Apr 18. PMID 16621868
- [Background] Taneva E, Borucki K, Wiens L, Makarova R, Schmidt-Lucke C, Luley C, Westphal S. Early effects on endothelial function of atorvastatin 40 mg twice daily and its withdrawal. Am J Cardiol. 2006 Apr 1;97(7):1002-6. doi: 10.1016/j.amjcard.2005.10.032. Epub 2006 Feb 13. PMID 16563905
- [Background] Kougias P, Chai H, Lin PH, Yao Q, Lumsden AB, Chen C. Effects of adipocyte-derived cytokines on endothelial functions: implication of vascular disease. J Surg Res. 2005 Jun 1;126(1):121-9. doi: 10.1016/j.jss.2004.12.023. PMID 15916985
- [Background] Mahmud A, Feely J. Adiponectin and arterial stiffness. Am J Hypertens. 2005 Dec;18(12 Pt 1):1543-8. doi: 10.1016/j.amjhyper.2005.06.014. PMID 16364823
- [Background] Ekmekci H, Ekmekci OB. The role of adiponectin in atherosclerosis and thrombosis. Clin Appl Thromb Hemost. 2006 Apr;12(2):163-8. doi: 10.1177/107602960601200203. PMID 16708117
- [Background] Nagasawa A, Fukui K, Kojima M, Kishida K, Maeda N, Nagaretani H, Hibuse T, Nishizawa H, Kihara S, Waki M, Takamatsu K, Funahashi T, Matsuzawa Y. Divergent effects of soy protein diet on the expression of adipocytokines. Biochem Biophys Res Commun. 2003 Nov 28;311(4):909-14. doi: 10.1016/j.bbrc.2003.10.087. PMID 14623267
- [Background] Qi L, Rimm E, Liu S, Rifai N, Hu FB. Dietary glycemic index, glycemic load, cereal fiber, and plasma adiponectin concentration in diabetic men. Diabetes Care. 2005 May;28(5):1022-8. doi: 10.2337/diacare.28.5.1022. PMID 15855561
- [Background] Polson DA, Thompson MP. Macronutrient composition of the diet differentially affects leptin and adiponutrin mRNA expression in response to meal feeding. J Nutr Biochem. 2004 Apr;15(4):242-6. doi: 10.1016/j.jnutbio.2003.11.009. PMID 15068818
- [Background] Rossi AS, Lombardo YB, Lacorte JM, Chicco AG, Rouault C, Slama G, Rizkalla SW. Dietary fish oil positively regulates plasma leptin and adiponectin levels in sucrose-fed, insulin-resistant rats. Am J Physiol Regul Integr Comp Physiol. 2005 Aug;289(2):R486-R494. doi: 10.1152/ajpregu.00846.2004. PMID 16014450
- [Background] Flachs P, Mohamed-Ali V, Horakova O, Rossmeisl M, Hosseinzadeh-Attar MJ, Hensler M, Ruzickova J, Kopecky J. Polyunsaturated fatty acids of marine origin induce adiponectin in mice fed a high-fat diet. Diabetologia. 2006 Feb;49(2):394-7. doi: 10.1007/s00125-005-0053-y. Epub 2006 Jan 6. PMID 16397791
- [Background] Chan LL, Chen Q, Go AG, Lam EK, Li ET. Reduced adiposity in bitter melon (Momordica charantia)-fed rats is associated with increased lipid oxidative enzyme activities and uncoupling protein expression. J Nutr. 2005 Nov;135(11):2517-23. doi: 10.1093/jn/135.11.2517. PMID 16251604
- [Background] Fisher FM, Trujillo ME, Hanif W, Barnett AH, McTernan PG, Scherer PE, Kumar S. Serum high molecular weight complex of adiponectin correlates better with glucose tolerance than total serum adiponectin in Indo-Asian males. Diabetologia. 2005 Jun;48(6):1084-7. doi: 10.1007/s00125-005-1758-7. Epub 2005 May 19. PMID 15902402
- [Background] Lara-Castro C, Luo N, Wallace P, Klein RL, Garvey WT. Adiponectin multimeric complexes and the metabolic syndrome trait cluster. Diabetes. 2006 Jan;55(1):249-59. PMID 16380500
- [Background] Sumpio BE, Riley JT, Dardik A. Cells in focus: endothelial cell. Int J Biochem Cell Biol. 2002 Dec;34(12):1508-12. doi: 10.1016/s1357-2725(02)00075-4. PMID 12379270
- [Background] Pearson JD. Normal endothelial cell function. Lupus. 2000;9(3):183-8. doi: 10.1191/096120300678828299. PMID 10805485
- [Background] Constans J, Conri C. Circulating markers of endothelial function in cardiovascular disease. Clin Chim Acta. 2006 Jun;368(1-2):33-47. doi: 10.1016/j.cca.2005.12.030. Epub 2006 Mar 10. PMID 16530177
- [Background] Tang Y, Lu A, Aronow BJ, Sharp FR. Blood genomic responses differ after stroke, seizures, hypoglycemia, and hypoxia: blood genomic fingerprints of disease. Ann Neurol. 2001 Dec;50(6):699-707. doi: 10.1002/ana.10042. PMID 11761467
- [Background] Cooney CA, Dave AA, Wolff GL. Maternal methyl supplements in mice affect epigenetic variation and DNA methylation of offspring. J Nutr. 2002 Aug;132(8 Suppl):2393S-2400S. doi: 10.1093/jn/132.8.2393S. PMID 12163699
- [Background] Jaenisch R, Bird A. Epigenetic regulation of gene expression: how the genome integrates intrinsic and environmental signals. Nat Genet. 2003 Mar;33 Suppl:245-54. doi: 10.1038/ng1089. PMID 12610534
- [Background] Rodenhiser D, Mann M. Epigenetics and human disease: translating basic biology into clinical applications. CMAJ. 2006 Jan 31;174(3):341-8. doi: 10.1503/cmaj.050774. PMID 16446478
- [Background] Sing CF, Stengard JH, Kardia SL. Genes, environment, and cardiovascular disease. Arterioscler Thromb Vasc Biol. 2003 Jul 1;23(7):1190-6. doi: 10.1161/01.ATV.0000075081.51227.86. Epub 2003 May 1. PMID 12730090
- [Background] Rakyan VK, Preis J, Morgan HD, Whitelaw E. The marks, mechanisms and memory of epigenetic states in mammals. Biochem J. 2001 May 15;356(Pt 1):1-10. doi: 10.1042/0264-6021:3560001. PMID 11336630
- [Background] Waterland RA, Lin JR, Smith CA, Jirtle RL. Post-weaning diet affects genomic imprinting at the insulin-like growth factor 2 (Igf2) locus. Hum Mol Genet. 2006 Mar 1;15(5):705-16. doi: 10.1093/hmg/ddi484. Epub 2006 Jan 18. PMID 16421170
- [Background] Esteller M, Almouzni G. How epigenetics integrates nuclear functions. Workshop on epigenetics and chromatin: transcriptional regulation and beyond. EMBO Rep. 2005 Jul;6(7):624-8. doi: 10.1038/sj.embor.7400456. PMID 15976819
- [Background] Dolinoy DC, Weidman JR, Waterland RA, Jirtle RL. Maternal genistein alters coat color and protects Avy mouse offspring from obesity by modifying the fetal epigenome. Environ Health Perspect. 2006 Apr;114(4):567-72. doi: 10.1289/ehp.8700. PMID 16581547
- [Background] Lorenz RL, Uedelhoven WM, Fischer S, Ruetzel A, Weber PC. A critical evaluation of urinary immunoreactive thromboxane: feasibility of its determination as a potential vascular risk indicator. Biochim Biophys Acta. 1989 Dec 8;993(2-3):259-65. doi: 10.1016/0304-4165(89)90174-8. PMID 2597697
- [Background] Nestel P, Fujii A, Zhang L. An isoflavone metabolite reduces arterial stiffness and blood pressure in overweight men and postmenopausal women. Atherosclerosis. 2007 May;192(1):184-9. doi: 10.1016/j.atherosclerosis.2006.04.033. Epub 2006 May 30. PMID 16730732